CLINICAL TRIAL: NCT04360213
Title: Advanced Multimodal Wireless Vital Signs Monitoring for Patients With Asthma and Anaphylaxis
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Shuai (Steve) Xu, Principal Investigator, Northwestern University
Other Study IDs: 2020-3403
Record Dates: First submitted 2020-04-15; First posted 2020-04-24 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Asthma in Children; Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children with Asthma: 1. Patients ages 1 to 17 years old
  2. Patients in the Emergency Department or admitted to the hospital for asthma exacerbation.
  Interventions: Device: Advanced multimodal wireless vital signs monitor
- Children with allergy: 1. Patients ages 1 to 17 years old
  2. Patients scheduled to do an oral food challenge
  Interventions: Device: Advanced multimodal wireless vital signs monitor

INTERVENTIONS:
Device: Advanced multimodal wireless vital signs monitor — Investigators have developed a lightweight, stretchable 'skin-like' membranes, called skin sensors. These small, paper-thin monitors were created by matching the mechanical properties of skin, and can be applied to the skin's surface without skin disturbance. Each patch is encapsulated using medical grade materials and applied using single use medical grade skin adhesive integrated with eco-fused fabric (moisture wicking layer between adhesives). The adhesive may be changed between uses, and the device itself can be cleaned with Super Sani-Cloth®, commonly used in the hospital setting.

SUMMARY:
The primary objective of this study is to assess the function and reliability of a non-invasive, skin-like electronic sensor.

We hypothesize that this skin sensor will address an unmet need to wirelessly, noninvasively, and rapidly assess critical vital signs and other measures essential to healthcare monitoring for patients with asthma and anaphylaxis.

DETAILED DESCRIPTION:
In clinical and home settings sensors to monitor vital parameters (including heart rate, ECG, respiratory rate, temperature, and pulse oximetry) require the application and removal of multiple, often bulky apparatuses. Furthermore, each requires constant, wired attachment to a power supply and operators, which can limit visibility and impair the ability to move a patient without interference. Serial measurements require significant time, as several devices with separate leads are applied and removed to obtain measurements. Due to the varying and often large measurement heads of different devices, readings may not be obtained at exactly the same skin location, which impairs comparability of serial measurements. Additionally, the process of measurement can disturb the skin area being measured.

Asthma and anaphylaxis are common entities in children. During exacerbations, frequent monitoring of the vital parameters described is necessary to guide medical decision-making. Asthma exacerbations are associated with mild to severe symptoms that include cough, wheeze, tachypnea, retractions, labored breathing and respiratory fatigue. Food allergy reactions are potentially severe with life-threatening symptoms of anaphylactic shock that include, choking, respiratory distress and loss of consciousness. In the most severe cases reactions can be fatal or require emergency and intensive care treatment in the hospital. Convenient, easy to use, vital signs monitors are especially important in pediatric populations as children have less ability to self-monitor or describe their physical symptoms of life-threatening anaphylaxis or asthma exacerbation.

The wearable sensors offer a new, non-invasive and easy to use way to monitor vital signs of patients with asthma and anaphylaxis. Our previous experience testing our wearable vital sign sensors in multiple pediatric and neonatal studies since 2016, have shown a strong correlation to existing standard of care monitor data outputs. Additionally, the sensors have received positive feedback from patients and physicians, on their comfort, ease of use, and application.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ages 1 to 17 years old
2. Patients scheduled to do an oral food challenge or managed in the ED or admitted to the hospital for asthma exacerbation.
3. For exploratory analyses of breath sounds, patients in the ED with signs and symptoms of lower respiratory tract infection (e.g., bronchiolitis, pneumonitis, pneumonia).

Exclusion Criteria

1. Patient's with fragile skin or skin conditions that would prevent them from having a sensor placed (including wounds, blistering, cracked or peeling skin, burns or skin that is bandaged/covered)

Ages: 1 Year to 17 Years | Sex: All
Age Groups: Child
Study Population: Children scheduled to come to the hospital or admitted into Emergency Department for allergy testing, anaphylaxis or asthma exacerbations.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Percent agreement with pilot sensor and current standard | 2 years

SECONDARY OUTCOMES:
Capture of patient feedback examining opinions on use of wearable sensors compared to standard of care devices.(Allergy patients) | 2 years
  Use of Standardized survey instrument: IRB 2020-3403 Allergy Survey 2.21.20 Collects data on users perceived value of wireless monitoring, comfort, application and ease of use.
Capture of patient feedback examining opinions on use of wearable sensors compared to standard of care devices.(Asthma patients) | 2 years
  Use of Standardized survey instrument: IRB 2020-3403 Asthma Survey 2.21.20 Collects data on users perceived value of wireless monitoring, comfort, application and ease of use.

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States